CLINICAL TRIAL: NCT03384043
Title: Using Smartphone Personal Assistant Technology to Improve Prospective Memory in Alzheimer's Disease
Brief Title: Comparing Smartphone Technology and a Memory Strategy on Improving Prospective Memory in Alzheimer's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Michael Scullin, Assistant Professor of Psychology and Neuroscience, Baylor University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 017-327; 1R21AG053161-01A1 (NIH)
Record Dates: First submitted 2017-12-18; First posted 2017-12-27 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: Alzheimer Disease; Cognitive Impairment, Mild; Dementia, Mild
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction; Dementia; Lymphoma, Follicular

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Smartphone Personal Assistant (Experimental): Participants will use the personal assistant feature of the smartphone ("Cortana") to provide reminders to perform prospective memory tasks at the appropriate time and location. In the current study, participants will press a button and verbally state "Cortana, I need to remember to..." for time--based tasks ("...take my medicine at 7pm") and event--based tasks ("pick-up milk at the grocery store).
  Interventions: Behavioral: Smartphone Personal Assistant
- Implementation Intention (Active Comparator): The implementation intention is a memory strategy, in which individuals verbally state when/where they will perform a prospective memory intention. In the current study, participants will verbally specify an external cue in a "When…then" format and record doing so using the smartphone's voice recorder app. They will use the implementation intention strategy for time--based tasks ("When it is 7pm, then I will remember to take my medicine"), and event--based tasks ("When I am at the grocery store, then I will remember to pick--up milk).
  Interventions: Behavioral: Implementation Intention

INTERVENTIONS:
Behavioral: Smartphone Personal Assistant — Electronic memory aids (e.g., pagers) are known to support memory for goals and intentions (prospective memory) in individuals with cognitive impairment. Smartphone technology has the potential to enhance the benefits of previous electronic memory aids because they can provide reminders not only at the correct time, but also at the correct location.
  Arms: Smartphone Personal Assistant
Behavioral: Implementation Intention — Verbally specifying when and where one intends to complete a goal or action (prospective memory) is known to improve the likelihood of later completing that prospective memory. The implementation intention is the best known memory strategy for prospective memory in patients with mild cognitive impairment.
  Arms: Implementation Intention

SUMMARY:
Alzheimer's disease is a debilitating condition for patients and their caregivers marked by hallmark cognitive symptoms (e.g., memory loss) as well as an impact on quality of life. Researchers and clinicians are learning that a specific type of memory, called prospective memory, may be particularly affected in mild Alzheimer's disease. Prospective memory is memory for future intentions, goals, and chores, and the loss of the neurocognitive processes supporting prospective memory may reduce independent functioning (e.g., medication adherence). The current study investigates a technology-based intervention to assist participants with their daily prospective memory tasks. Participants with mild cognitive impairment and mild Alzheimer's disease will be trained to use a smartphone for four weeks. Smartphone acceptability, usability, and overall user experience will be measured. Furthermore, participants will be tested on completion of daily prospective memory tasks. In one group, participants will train to use the smartphone personal assistant reminder system, which reminds participants of their goals, tasks, and chores at the appropriate time or location. In a comparison group, participants will also carry a smartphone but will train to use a memory strategy in which they verbalize external cues to remind them to perform their goals, tasks, and chores. The goal of this research is to inform whether smartphone technology or a memory strategy can be used to reduce memory burden and improve daily, independent functioning in participants with mild Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MCI or dementia at a neurology and/or neuropsychology office visit in the BSWH Temple region, or neuropsychology office visit in the RR BSWH region within 12 months of the study contact (Specific ICD Codes outlined below).
* Interest in participating in research
* Able and willing to bring a legally authorized representative (spouse or medical power of attorney) to initial training session.
* Able to independently consent according to the results of a structured capacity to consent interview OR is interested after going through the consent process but does not pass capacity to consent inventory AND has a legally authorized representative available to provide proxy consent.
* Presence of no more than mild dementia on the basis of telephone administered cognitive screening instrument (TICS-M) & Collateral/Informant ADL Measure

  o Using the TICS-M and published normative data, all subjects must have scores that are around -1 to -2 standard deviations for demographically corrected norms (National Institute of Aging-Alzheimer's Association recommended criteria for the very mild to mild stages of Alzheimer's disease; Albert et al., 2011; McKhann et al., 2011).
* Etiology of the dementia or MCI can be varied or unknown at the time of the screening criteria.

Exclusion Criteria:

* Presence of severe cognitive impairment defined by a TICS-M score <-2 standard deviations from the mean.
* Semi-structured telephone clinical interview and/or chart review suggest:

  * Serious mental illness (schizophrenia, bipolar, or depression with suicidal ideation in the last 30 days) are present and significantly contributing to the current presentation
  * Uncorrected hearing loss, visual loss, or motoric dysfunction would preclude using the smartphone.
* English language proficiency (whether due to English as a second language or the presence of aphasia) significantly interferes with completion of telephone screening procedures or would be clinically suspected to interfere with completion of the study process.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Objective Prospective Memory Performance | Measured for 4 weeks.
  Performance on the experimenter-assigned time-based and event-based prospective memory tasks (number of tasks completed).

SECONDARY OUTCOMES:
Quality of Life - Positive Affect and Well-Being | Pre-Intervention and Post-Intervention (4 weeks)
  Participants will complete the Quality of Life in Neurological Disorders (Neuro-QOL) subscale titled "Positive Affect and Well-Being." This subscale has 9 items that are rated from Never to Always. The subscale total scores range from 9 (minimum) to 45 (maximum), with higher scores indicating better outcomes
Quality of Life - Ability to Participate in Social Roles and Activities | Pre-Intervention and Post-Intervention (4 weeks)
  Participants will complete the Quality of Life in Neurological Disorders (Neuro-QOL) subscale titled "Ability to Participate in Social Roles and Activities." This subscale has 8 items that are rated from Never to Always. The subscale total scores range from 8 (minimum) to 40 (maximum), with higher scores indicating better outcomes.
Quality of Life - Satisfaction with Social Roles and Activities | Pre-Intervention and Post-Intervention (4 weeks)
  Participants will complete the Quality of Life in Neurological Disorders (Neuro-QOL) subscale titled "Satisfaction with Social Roles and Activities." This subscale has 8 items that are rated from Not at All to Very Much. The subscale total scores range from 8 (minimum) to 40 (maximum), with higher scores indicating better outcomes.
Quality of Life - Cognitive Function | Pre-Intervention and Post-Intervention (4 weeks)
  Participants will complete the Quality of Life in Neurological Disorders (Neuro-QOL) subscale titled "Cognitive Function." This subscale has 8 items. The first four items are rated from Never to Very Often, and the last four items are rated from No Difficulty to Cannot Do. The subscale total scores range from 8 (minimum) to 40 (maximum), with higher scores indicating better outcomes.
Subjective Memory Performance Questionnaire | Pre-Intervention and Post-Intervention (4 weeks)
  The Prospective and Retrospective Memory Questionnaire uses a 5-point scale to assess the frequency of retrospective and prospective memory failures such as forgetting to take a pill.
Perceived Memory Structured Interview | Pre-Intervention and Post-Intervention (4 weeks)
  The experimenter will conduct a structured interview session at baseline to determine participants' most important, common, and challenging prospective memory tasks. At follow-up, participants will rate whether each memory issue described at baseline was much worse (1), worse (2), normal (3), better (4), or much better (5) than usual over the last month.
Use of Technology/Strategy | Measured for 4 weeks
  The number of times the personal assistant feature and voice-recorder system were used.
Instrumental Activities of Daily Living | Pre-Intervention and Post-Intervention (4 weeks)
  Scale on participants' ability to complete instrumental activities of daily living, such as housekeeping, financing, and medication activities.
Smartphone Acceptability/Usability Scale | Pre-Intervention and Post-Intervention (4 weeks)
  Scale to assess the acceptability and usability of the smartphone (Ben Zeev et al., 2014). The scale includes 26 items to which participants respond agree, neutral, or disagree, with agree indicating the favorable outcome on 21 items, and disagree indicating the favorable outcome on 5 items.
Training Duration | Pre-Intervention
  Number of minutes to complete smartphone training

CONTACTS AND LOCATIONS:
Overall Officials: Michael Scullin, PhD, Principal Investigator — Baylor University
Locations (1):
- Baylor Scott & White Medical Center, Temple, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided
De-identified data will be shared with any interested researcher who adheres to Health Insurance Portability and Accountability Act (HIPAA) requirements.

REFERENCES:
- [Background] Ben-Zeev D, Brenner CJ, Begale M, Duffecy J, Mohr DC, Mueser KT. Feasibility, acceptability, and preliminary efficacy of a smartphone intervention for schizophrenia. Schizophr Bull. 2014 Nov;40(6):1244-53. doi: 10.1093/schbul/sbu033. Epub 2014 Mar 8. PMID 24609454